CLINICAL TRIAL: NCT06815861
Title: Perioperative Morbidity in Adult Scoliotic Surgery: Analysis of a Series From Brest
Brief Title: Perioperative Morbidity in Adult Scoliotic Surgery: Analysis of a Series From Brest (MOSCA-B)
Acronym: MOSCA-B
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0313 - MOSCA-B
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-10

CONDITIONS: Adult Scoliosis; Spine Deformity; Neurosurgery
Keywords: adult scoliosis; spine deformity; neurosurgery; spine surgery
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scoliosis surgery is an invasive procedure essential for alleviating significant pain and improving the physical, psychological, aesthetic, professional, and social well-being of patients. However, it carries a considerable risk of perioperative complications. This retrospective study, conducted at Brest University Hospital since 2017, aims to analyze these complications to provide a detailed assessment, particularly since the introduction of the OARM (intraoperative CT navigation), with the goal of optimizing the safety and effectiveness of surgical interventions. The complications studied include neurological, infectious, mechanical, and cardiopulmonary complications, along with an additional "other" category for rare complications. The period analyzed extends from the immediate postoperative phase to the most recent follow-up consultation with the referring surgeon, which varies depending on the duration of follow-up for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient affiliated with a social security system
* Who underwent scoliosis surgery between 2017 and 2024 at the Brest University Hospital

Exclusion Criteria:

Patients under legal protection (guardianship, curatorship, etc.) Refusal to participate (expressed opposition) History of scoliosis surgery performed by another surgeon, regardless of the center or year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient Who underwent scoliosis surgery between 2017 and 2024 at the Brest University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of postoperative complications | at the time of inclusion
  Number of complications (raw description), followed by univariate analysis to exclude confounding factors

SECONDARY OUTCOMES:
ODI SORE | at the time of inclusion
  ODI SCORE after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement